CLINICAL TRIAL: NCT06959459
Title: Evaluation of the Safety and Efficacy of Artificial Bone Repair Materials for Repair of Long Bone Defects in the Extremities: A Prospective, Randomized Controlled, Single-Blind, Non-Inferiority Clinical Trial
Brief Title: Evaluation of the Safety and Efficacy of Artificial Bone Repair Materials for Repair of Long Bone Defects in the Extremities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhang Wei, Deputy head of orthopedics, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024QX008-KS002
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Bone Defects of the Limbs

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Use of artificial bone repair materials produced by Changzhou Bone-Renewal Medical Technologies LLC.
  Interventions: Device: Intervention Group:Use of artificial bone repair materials produced by Changzhou Bone-Renewal Medical Technologies LLC.
- Control group (Active Comparator): Use of β-tricalcium phosphate bioceramics produced by Shanghai Biolu Biomaterials Co., Ltd.
  Interventions: Device: Control group: Use of β-tricalcium phosphate bioceramics produced by Shanghai Biolu Biomaterials Co., Ltd.

INTERVENTIONS:
Device: Intervention Group:Use of artificial bone repair materials produced by Changzhou Bone-Renewal Medical Technologies LLC. — Use of artificial bone repair materials produced by Changzhou Bone-Renewal Medical Technologies LLC.
  Arms: Intervention Group
Device: Control group: Use of β-tricalcium phosphate bioceramics produced by Shanghai Biolu Biomaterials Co., Ltd. — Use of β-tricalcium phosphate bioceramics produced by Shanghai Biolu Biomaterials Co., Ltd.
  Arms: Control group

SUMMARY:
Evaluation of the Safety and Efficacy of Artificial Bone Repair Materials for Repair of Long Bone Defects in the Extremities: A Prospective, Randomized Controlled, Single-Blind, Non-Inferiority Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 60 years old, regardless of sex;
2. Cavitary bone defects in the limbs requiring bone grafting treatment;
3. Bone defect volume ≥ 1 cm³ and ≤ 8 cm³, with only one bone defect requiring intervention;
4. Subjects or their legal guardians can understand the study objectives, demonstrate sufficient compliance with the study protocol, and sign the informed consent form.

Exclusion Criteria:

1. Open fractures with wound contamination;
2. Repair of infectious bone defects;
3. Structural bone grafting required at the defect site;
4. Osteofascial compartment syndrome in the affected limb scheduled for surgery;
5. Presence of systemic infection, uncontrolled local infection at the surgical site, malignant tumor (including metastatic tumors) at the defect site, osteonecrosis at the defect site, severe nerve/soft tissue/vascular injury at the defect site, confirmed severe malnutrition, or dysfunction/failure of other vital organs;
6. Calcium and phosphorus metabolic abnormalities (calcium/phosphorus levels > 1.5 times the upper limit of normal values);
7. History of diabetes with fasting blood glucose ≥ 6.1 mmol/L;
8. Coagulation dysfunction (prothrombin time [PT] or activated partial thromboplastin time [APTT] > 2 times the upper limit of normal values);
9. Use of chemotherapeutic agents or receipt of radiotherapy within 3 months prior to enrollment;
10. Cumulative use of corticosteroids or growth factors for ≥ 14 days within 1 month prior to enrollment;
11. Long-term use of sedative-hypnotic drugs (continuous use for > 3 months) or non-steroidal anti-inflammatory drugs (NSAIDs, continuous use for > 3 months);
12. Known allergy to bovine-derived materials or collagen products;
13. Pregnant or lactating females;
14. Participation in other interventional clinical trials for drugs or medical devices within 1 month prior to enrollment;
15. Any other conditions where investigators, in their professional judgment, deem the subject ineligible to participate in the trial for the subject's safety or benefit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Bone graft fusion rate | 24weeks after surgery

SECONDARY OUTCOMES:
Bone defect healing rate | 4 and 12 weeks after surgery
New bone formation rate | 4, 12 and 24 weeks after surgery
SF-36 scale | 24 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hosptial, Beijing, China

IPD SHARING:
Plan to Share IPD: No